CLINICAL TRIAL: NCT02200913
Title: Effects of Core Stabilization Exercise on Balance in Low Back Pain Patients With Clinical Lumbar Instability
Brief Title: Effects of Core Stabilization Exercise on Balance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Wantanee Yodchaisarn, Research Center in Back, Neck, Other Joint Pain and Human Performance, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WYodchaisarn
Record Dates: First submitted 2014-07-24; First posted 2014-07-25 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Lumbar Spine Instability

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- core stabilization exercise (Experimental): core stabilization exercise 2 times/week 10 weeks
  Interventions: Other: general trunk strengthening exercise
- general trunk strengthening exercise (Experimental): general trunk strengthening exercise, 2 times/week, 10 weeks
  Interventions: Other: core stabilization exercise

INTERVENTIONS:
Other: core stabilization exercise — core stabilization exercise, 2 times/week, 10 weeks
  Arms: general trunk strengthening exercise
Other: general trunk strengthening exercise — general trunk strengthening exercise, 2 times/week, 10 weeks
  Arms: core stabilization exercise

SUMMARY:
Recent studies indicate that patients with chronic low back pain (LBP) present problems in balance. Alterations in proprioception are the possible causes of alteration of postural balance in LBP.

Previous studies reported an improvement of CSE on joint mobility, pain, functional disability, and trunk muscle activation pattern in patients with clinical lumbar instability (CLI); however, it was an immediate effect. However, previous studies did not report indirect effect may occur in CLI as postural balance and other kinds of exercise as strengthening in CLI. The general trunk strengthening exercise is common used in physical therapy clinic on LBP, that improve pain, physical disability, and trunk muscles activity. To our knowledge, the usefulness of CSE has not yet been investigated in CLI patients with outcome measure of balance.

The present study will conduct to fill the gaps of previous studies which will provide immediate-, accumulative- and detraining-effects of CSE on postural balance, pain intensity and ratio activation of trunk muscles and included blinding process of the assessor.

DETAILED DESCRIPTION:
Low back pain (LBP) is the most common musculoskeletal complaint. In most LBPs, it is benign and disappears within six weeks, but approximately 20% of individuals with LBP do not show any improvement in their condition, which may progress to chronic low back pain. LBP not only interferes with biomechanical change, but also causes ability to work leading to reduced productivity, economic burden to individuals and society for medical costs Recent studies indicate that patients with chronic low back pain present diminished postural control, manifesting problems in balance. Postural balance is controlled by sensory information, central processing and neuromuscular responses. Alterations in proprioception are the possible causes of alteration of postural balance in individuals with low back pain.

For clinical studies using core stabilization exercise (CSE) as treatment have revealed conflicting findings on pain, functional disability and muscle responses in chronic LBP. The few studies that investigated CSE as an isolated factor. Kumar (2011) reported an improvement of CSE on joint mobility and pain pressure threshold in patients with clinical lumbar instability; however, it was an immediate effect of CSE and blinding process was not performed. However, an effectiveness of CSE on pain intensity, functional disability, and trunk muscle activation pattern were improved in clinical lumbar instability (CLI). In addition, after 10-week CSE provides greater training and retention effects on pain-related outcomes and induced activation of deep abdominal muscles in CLI compared with conventional treatment (stretching exercise and hot pack). However, previous studies did not report indirect effect may occur in CLI as postural balance and other kinds of exercise as strengthening in CLI. The general trunk strengthening exercise is common used in physical therapy clinic on LBP, that improve pain, physical disability, and trunk muscles activity. To our knowledge, the usefulness of CSE technique as abdominal drawing-in maneuver (ADIM) has not yet been investigated in CLI patients with outcome measure of balance.

ELIGIBILITY:
Inclusion Criteria:

* male or female
* aged between 20-60 years
* low back pain (LBP) with or without radiating leg pain for period of at least 12 weeks
* answer 'yes' at least seven items of questionnaire
* present positive sign of the aberrant movement sign
* Present at least one positive sign from painful catch , prone instability catch test, or apprehension symptom

Exclusion Criteria:

* Be pregnant.
* Have serious spinal pathology: spinal fracture, spinal malignancy or spinal infection
* Have quada equina syndrome
* Have neurological deficit (at least 2 of the following signs: weakness of lower limbs (muscle power < grade 3 using manual muscle test), reflex changes, or abnormality or loss of sensation of lower limbs associated with the spinal nerve root
* Have obvious abnormal movement of the lumbar motion segment when assessed by flexion-extension radiographs: sagittal plane translation larger than 4.5mm or 15 percent of vertebral body width according to other vertebral segment, or sagittal plane rotation larger than 15 degrees at L1-L2, L2-L3 or L3-L4, 20 degrees at L4-L5 or 25 degrees at L5-S1
* Have visual disorder, vestibular disorder, neuromuscular diseases such as polyneuropathy, or diabetes neuropathy
* Participate in their intervention less than 5 out of the 10 week of intervention.
* Regularly treat with core stabilization exercise (CSE), or trunk strengthen exercises.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
center of pressure | up to 3-months after the last intervention session

CONTACTS AND LOCATIONS:
Overall Officials: Wantanee Yodchaisarn, M.Sc., Principal Investigator — Research Center in Back, Neck, Other Joint Pain and Human Performance, Khon Kaen University
Locations (1):
- Research Center in Back, Neck, Other Joint Pain and Human Performance, Khon Kaen, Thailand

REFERENCES:
- [Result] Puntumetakul R, Areeudomwong P, Emasithi A, Yamauchi J. Effect of 10-week core stabilization exercise training and detraining on pain-related outcomes in patients with clinical lumbar instability. Patient Prefer Adherence. 2013 Nov 19;7:1189-99. doi: 10.2147/PPA.S50436. eCollection 2013. PMID 24399870